CLINICAL TRIAL: NCT02564926
Title: Effects of Dapagliflozin Compared With Glimepiride on Body Composition in Patients With Type 2 Diabetes Inadequately Controlled With Metformin
Brief Title: Foxiga Korea Local Phase 4 Study
Acronym: BEYOND
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D1690L00067
Record Dates: First submitted 2015-09-23; First posted 2015-10-01 (Estimated); Results first posted 2019-08-20 (Actual); Last update posted 2019-08-20 (Actual); Status verified 2019-08

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: DM
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — dapagliflozin; glimepiride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Dapagliflozin (Experimental): Dapagliflozin 10mg + Metformin 1000mg
  Interventions: Drug: Dapagliflozin
- Glimepiride (Active Comparator): Glimepiriide 1-2mg + Metformin 1000mg
  Interventions: Drug: Glimepiride

INTERVENTIONS:
Drug: Dapagliflozin — Subject who will be randomized to the 'Dapagliflozin arm' will be treated with dapagliflozin 10mg + Metformin 1000 mg as Diabetes Treatment
  Arms: Dapagliflozin
Drug: Glimepiride — Subject who will be randomized to the 'Glimepiride arm' will be treated with glimepiride 1-2mg + Metformin 1000 mg as Diabetes Treatment
  Arms: Glimepiride

SUMMARY:
To evaluate the effect of dapagliflozin on body composition in Korean T2DM subjects.12-month, randomised, open-label, parallel-group, multi-centre phase IV study.

DETAILED DESCRIPTION:
This is a 52 weeks, randomized, open-label, parallel-group, multi-centres phase IV study.

Participants will be randomized 1:1 to receive dapagliflozin 10 mg qd or glimepiride 1~2 mgqd in an open-label manner for 12 months as add-on to metformin 1000 mg.

Parallel group study design was chosen. In order maintain the practicality of the phase IV study, open label design of study drug delivery was chosen. The reading of the DXA scans will be conducted by one expert in blinded manner. Glimepiride is the most frequently used SUs in Korea and therefore this was chosen as comparator.Dapagliflozin treatment will be associated with reduction of total body FM, BW, abdominal VAT and SAT volume compared with glimepiride.

ELIGIBILITY:
Inclusion Criteria:

1. Adults with T2DM (Male or female, ≥ 19 and ≤ 75 yrs)
2. Patients in insufficient glycemic control (HbA1c > 7.5% and < 9.5% in recent 4 weeks)
3. Patients with an unchanged dose of metformin (≥ 1,000 mg/day) for > 8 weeks prior to randomization
4. Written informed consent
5. WOCBP must take precautions to avoid pregnancy throughout the study and for 4 weeks after intake of the last dose.

   * WOCBP must have a negative urine pregnancy test at screening visit WOCBP include any female who has experienced menarche and who has not undergone successful surgical sterilization (hysterectomy, bilateral tubal ligation or bilateral oophorectomy) or is not postmenopausal.
   * WOCBP must be willing to use a medically accepted method of contraception that is considered reliable in the judgment of the Investigator.

Exclusion Criteria:

1. Type 1 diabetes or history of diabetic ketoacidosis
2. Pregnant or breast-feeding patients
3. eGFR < 60 mL/min/1.73 m2 (MDRD) on visit 1.
4. Indication of active liver disease (AST/ALT/total bilirubin > 3 X upper limits of normal) on visit 1.
5. Acute coronary syndrome, stroke or TIA within 3 months prior to randomization
6. Bariatric surgery within 2 years; treatment of anti-obesity drugs 3 months prior to randomization; any treatment leading to unstable body weight. (Unstable body weight is considered reliable in the judgment of the Investigator.)
7. History of bladder cancer or history of radiation therapy to the lower abdomen or pelvis at any time
8. History of any other malignancy within 5 years (with the exception of successfully treated non-melanoma skin cancers)
9. History of alcohol or drug abuse judged by physician within 3 months prior to randomization
10. Concomitant participation in any other clinical study.

Ages: 19 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 125 (Actual)
Dates: Start 2016-01-05 (Actual); Primary Completion 2018-01-15 (Actual); Study Completion 2018-01-15 (Actual)

CONTACTS AND LOCATIONS:
Locations (11):
- South Korea (11):
  - Research Site, Ansan-si
  - Research Site, Changwon-si
  - Research Site, Daegu
  - Research Site, Daejeon
  - Research Site, Goyang-si
  - Research Site, Incheon
  - Research Site, Seongnam-si
  - Research Site, Seoul
  - Research Site, Suwon
  - Research Site, Uijeongbu-si
  - Research Site, Wŏnju

REFERENCES:
- See also: D1690l00067_CSP_Redacted — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=3942&filename=D1690l00067_CSP_Redacted.pdf
- See also: D1690l00067_SAP_Redacted — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=3942&filename=D1690l00067_SAP_Redacted.pdf

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First patient enrolled: 05 January 2016 Last patient last visit: 15 January 2018
Pre-assignment Details: 178 patients provided informed consent. 121 patients received study treatment and were included in the SAF population. 112 patients received study treatment and had at least one post-baseline primary efficacy assessment and were included in the FAS population (56 patients in each treatment group).
Period: Overall Study
Arm/Group | Dapagliflozin | Glimepiride
Started (121 patients received study treatment and were included in the SAF population.) | 60 | 61
Completed (Study Treatment/Entire Study Completed) | 52 | 54
Not Completed | 8 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Dapagliflozin | Glimepiride | Total
Number analyzed (Participants) | 60 | 61 | 121
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.6 (9.09) | 55.7 (10.24) | 55.2 (9.66)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 34 | 57
  Male | 37 | 27 | 64
Race/Ethnicity, Customized [Number; unit: Participants]
  Korean | 60 | 61 | 121

OUTCOME MEASURES:

1. Primary Outcome: Adjusted Mean Changes From Baseline in Total Body Fat Mass by DXA Scan
Description: Adjusted mean changes in total body fat mass from baseline using DXA scan in 52 weeks after the start of the treatment
Time Frame: From baseline to Week 52
Measure: Least Squares Mean (95% Confidence Interval); unit: grams
Arm/Group | Dapagliflozin | Glimepiride
Number analyzed (Participants) | 56 | 56
grams | -1485.69 [-2025.543 to -945.844] | 1096.34 [556.489 to 1636.187]
Statistical Analysis 1: Comparison: Dapagliflozin vs Glimepiride; Test type: Other; p < 0.001, ANCOVA; LS mean difference (kg) = -2.6, 95% CI 2-sided [-3.346 to -1.819]

2. Secondary Outcome: Adjusted Mean Change in HbA1c at Week 52
Description: Adjusted Mean Change in HbA1c at Week 52
Time Frame: From baseline to Week 52
Measure: Least Squares Mean (95% Confidence Interval); unit: percentages
Arm/Group | Dapagliflozin | Glimepiride
Number analyzed (Participants) | 56 | 56
percentages | -1.00 [-1.259 to -0.745] | -0.54 [-0.802 to -0.287]
Statistical Analysis 1: Comparison: Dapagliflozin vs Glimepiride; Test type: Other; p = 0.014, Mixed Models Analysis; LS mean difference (%) = -0.46, 95% CI 2-sided [-0.821 to -0.094]

3. Secondary Outcome: HbA1c <7.0% at Week 52
Description: HbA1c <7.0% at Week 52
Time Frame: 52 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Dapagliflozin | Glimepiride
Number analyzed (Participants) | 56 | 56
Participants
  Count of participants that achieved the response | 27 | 22
Statistical Analysis 1: Comparison: Dapagliflozin vs Glimepiride; Test type: Other; p = 0.343, Regression, Logistic; Odds Ratio (OR) = 1.45, 95% CI 2-sided [0.673 to 3.113]

4. Secondary Outcome: Adjusted Mean Change in Fasting Blood Sugar (FBS) at Week 52
Description: Adjusted Mean Change in Fasting Blood Sugar (FBS) at Week 52
Time Frame: From baseline to Week 52
Measure: Least Squares Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Dapagliflozin | Glimepiride
Number analyzed (Participants) | 56 | 56
mg/dL | -30.94 [-40.084 to -21.800] | -12.70 [-21.786 to -3.607]
Statistical Analysis 1: Comparison: Dapagliflozin vs Glimepiride; Test type: Other; p = 0.006, Mixed Models Analysis; LS mean difference (mg/dL) = -18.25, 95% CI 2-sided [-31.140 to -5.351]

5. Secondary Outcome: Adjusted Mean Change in Total Body Weight at Week 52
Description: Adjusted Mean Change in Total Body Weight at Week 52
Time Frame: From baseline to Week 52
Measure: Least Squares Mean (95% Confidence Interval); unit: kg
Arm/Group | Dapagliflozin | Glimepiride
Number analyzed (Participants) | 56 | 56
kg | -2.4 [-3.104 to -1.664] | 1.3 [0.545 to 1.984]
Statistical Analysis 1: Comparison: Dapagliflozin vs Glimepiride; Test type: Other; p < 0.001, Mixed Models Analysis; LS mean difference (kg) = -3.7, 95% CI 2-sided [-4.667 to -2.631]

6. Secondary Outcome: Adjusted Mean Change in Waist Circumference at Week 52
Description: Adjusted Mean Change in Waist Circumference at Week 52
Time Frame: From baseline to Week 52
Measure: Least Squares Mean (95% Confidence Interval); unit: cm
Arm/Group | Dapagliflozin | Glimepiride
Number analyzed (Participants) | 56 | 56
cm | -2.37 [-3.480 to -1.253] | -0.16 [-1.271 to 0.957]
Statistical Analysis 1: Comparison: Dapagliflozin vs Glimepiride; Test type: Other; p = 0.006, Mixed Models Analysis; LS mean difference (cm) = -2.21, 95% CI 2-sided [-3.785 to -0.635]

7. Secondary Outcome: Adjusted Mean Change in Body Mass Index (BMI) at Week 52
Description: Adjusted Mean Change in Body Mass Index (BMI) at Week 52
Time Frame: From baseline to Week 52
Measure: Least Squares Mean (95% Confidence Interval); unit: kg/m^2
Arm/Group | Dapagliflozin | Glimepiride
Number analyzed (Participants) | 56 | 56
kg/m^2 | -0.91 [-1.172 to -0.640] | 0.46 [0.194 to 0.726]
Statistical Analysis 1: Comparison: Dapagliflozin vs Glimepiride; Test type: Other; p < 0.001, Mixed Models Analysis; LS mean difference (kg/m2) = -1.37, 95% CI 2-sided [-1.742 to -0.990]

8. Secondary Outcome: Adjusted Mean Change in Systolic Blood Pressure (SBP) at Week 52
Description: Adjusted Mean Change in Systolic Blood Pressure (SBP) at Week 52
Time Frame: From baseline to Week 52
Measure: Least Squares Mean (95% Confidence Interval); unit: mmHg
Arm/Group | Dapagliflozin | Glimepiride
Number analyzed (Participants) | 56 | 56
mmHg | -2.18 [-5.123 to 0.766] | 4.63 [1.682 to 7.570]
Statistical Analysis 1: Comparison: Dapagliflozin vs Glimepiride; Test type: Other; p = 0.002, Mixed Models Analysis; LS mean difference (mmHg) = -6.81, 95% CI 2-sided [-10.969 to -2.641]

9. Secondary Outcome: Adjusted Mean Change in Diastolic Blood Pressure (DBP) at Week 52
Description: Adjusted Mean Change in Diastolic Blood Pressure (DBP) at Week 52
Time Frame: From baseline to Week 52
Measure: Least Squares Mean (95% Confidence Interval); unit: mmHg
Arm/Group | Dapagliflozin | Glimepiride
Number analyzed (Participants) | 56 | 56
mmHg | -0.25 [-2.523 to 2.023] | 2.36 [0.092 to 4.638]
Statistical Analysis 1: Comparison: Dapagliflozin vs Glimepiride; Test type: Other; p = 0.110, Mixed Models Analysis; LS mean difference (mmHg) = -2.61, 95% CI 2-sided [-5.829 to 0.600]

10. Secondary Outcome: Adjusted Mean Change in Visceral Adipose Tissue (VAT) Area at Week 52
Description: Adjusted Mean Change in Visceral Adipose Tissue (VAT) area at Week 52
Time Frame: From baseline to Week 52
Measure: Least Squares Mean (95% Confidence Interval); unit: cm^2
Arm/Group | Dapagliflozin | Glimepiride
Number analyzed (Participants) | 56 | 56
cm^2 | -16.06 [-23.806 to -8.317] | 1.48 [-6.407 to 9.377]
Statistical Analysis 1: Comparison: Dapagliflozin vs Glimepiride; Test type: Other; p = 0.002, ANCOVA; LS mean difference (cm2) = -17.55, 95% CI 2-sided [-28.603 to -6.489]

11. Secondary Outcome: Adjusted Mean Change in Subcutaneous Adipose Tissue (SAT) Area at Week 52
Description: Adjusted Mean Change in Subcutaneous Adipose Tissue (SAT) area at Week 52
Time Frame: From baseline to Week 52
Measure: Least Squares Mean (95% Confidence Interval); unit: cm^2
Arm/Group | Dapagliflozin | Glimepiride
Number analyzed (Participants) | 56 | 56
cm^2 | -5.41 [-11.804 to 0.994] | 12.98 [6.462 to 19.506]
Statistical Analysis 1: Comparison: Dapagliflozin vs Glimepiride; Test type: Other; p < 0.001, ANCOVA; LS mean difference (cm2) = -18.39, 95% CI 2-sided [-27.561 to -9.218]

12. Secondary Outcome: Adjusted Mean Change in Visceral to Subcutaneous Adipose Tissue Ratio at Week 52
Description: Adjusted Mean Change in Visceral to Subcutaneous Adipose Tissue Ratio at Week 52
Time Frame: From baseline to Week 52
Measure: Least Squares Mean (95% Confidence Interval); unit: ratio
Arm/Group | Dapagliflozin | Glimepiride
Number analyzed (Participants) | 56 | 56
ratio | -0.05 [-0.115 to 0.017] | -0.02 [-0.084 to 0.050]
Statistical Analysis 1: Comparison: Dapagliflozin vs Glimepiride; Test type: Other; p = 0.503, ANCOVA; LS mean difference = -0.03, 95% CI 2-sided [-0.127 to 0.063]

13. Secondary Outcome: Adjusted Mean Change in Lean Body Mass at Week 52
Description: Adjusted Mean Change in Lean Body Mass at Week 52
Time Frame: From baseline to Week 52
Measure: Least Squares Mean (95% Confidence Interval); unit: Kg
Arm/Group | Dapagliflozin | Glimepiride
Number analyzed (Participants) | 56 | 56
Kg | -1.1 [-1.608 to -0.570] | 0.2 [-0.329 to 0.683]
Statistical Analysis 1: Comparison: Dapagliflozin vs Glimepiride; Test type: Other; p < 0.001, ANCOVA; LS mean difference = -1.3, 95% CI 2-sided [-1.992 to -0.540]

14. Secondary Outcome: Adjusted Mean Change in Adinopectin at Week 52
Description: Adjusted Mean Change in Adinopectin at Week 52
Time Frame: From baseline to Week 52
Measure: Least Squares Mean (95% Confidence Interval); unit: ng/mL
Arm/Group | Dapagliflozin | Glimepiride
Number analyzed (Participants) | 56 | 56
ng/mL | 1746.66 [1296.144 to 2197.181] | 1088.95 [638.431 to 1539.468]
Statistical Analysis 1: Comparison: Dapagliflozin vs Glimepiride; Test type: Other; p = 0.044, ANCOVA; LS mean difference (ng/mL) = 657.71, 95% CI 2-sided [18.325 to 1297.101]

15. Secondary Outcome: Adjusted Mean Change in High Sensitivity C-Reactive Protein (hsCRP) at Week 52
Description: Adjusted Mean Change in High Sensitivity C-Reactive Protein (hsCRP) at Week 52
Time Frame: From baseline to Week 52
Measure: Least Squares Mean (95% Confidence Interval); unit: mg/L
Arm/Group | Dapagliflozin | Glimepiride
Number analyzed (Participants) | 56 | 56
mg/L | -0.51 [-1.030 to 0.014] | -0.39 [-0.914 to 0.131]
Statistical Analysis 1: Comparison: Dapagliflozin vs Glimepiride; Test type: Other; p = 0.756, ANCOVA; LS mean difference (mg/L) = -0.12, 95% CI 2-sided [-0.858 to 0.625]

16. Primary Outcome: Adjusted Mean Changes From Baseline in Percentage of Total Body Fat Assessed by DXA Scan
Description: Adjusted mean percent changes in total body fat mass from baseline using DXA scan in 52 weeks after the start of the treatment
Time Frame: From baseline to Week 52
Measure: Least Squares Mean (95% Confidence Interval); unit: percent change
Arm/Group | Dapagliflozin | Glimepiride
Number analyzed (Participants) | 56 | 56
percent change | -1.21 [-1.821 to -0.604] | 0.73 [0.123 to 1.341]
Statistical Analysis 1: Comparison: Dapagliflozin vs Glimepiride; Test type: Other; p < 0.001, ANCOVA; LS mean difference (%) = -1.94, 95% CI 2-sided [-2.807 to -1.082]

ADVERSE EVENTS:
Time Frame: 52 weeks
Arm/Group | Dapagliflozin | Glimepiride
All-Cause Mortality (participants affected / at risk) | 0/60 | 0/61
Serious Adverse Events (participants affected / at risk) | 6/60 | 6/61
Other Adverse Events (participants affected / at risk) | 11/60 | 10/61
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dapagliflozin (N=60) | Glimepiride (N=61)
Pyelonephritis acute (Infections and infestations) | 0 (0) | 1 (1)
Ankle fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Joint dislocation (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Rib fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Splenic injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Subdural haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Migraine (Nervous system disorders) | 0 (0) | 1 (1)
Transient ischaemic attack (Nervous system disorders) | 1 (1) | 0 (0)
Conversion disorder (Psychiatric disorders) | 1 (2) | 0 (0)
Trigeminal neuralgia (Nervous system disorders) | 0 (0) | 1 (1)
Tibia fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Chest pain (General disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dapagliflozin (N=60) | Glimepiride (N=61)
Toothache (Gastrointestinal disorders) | 4 (5) | 1 (1)
Nasopharyngitis (Infections and infestations) | 4 (4) | 2 (2)
Hypoglycaemia (Metabolism and nutrition disorders) | 3 (3) | 7 (12)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
* The Institution and PI shall provide the Company with copies of any materials relating to the Study that either intends to publish (or submit for publication) or make any presentations relating to, at least 30 days in advance of publication
* At the request of the Company, the Institution and PI shall withhold publication for a period of 90 days from the date on which the Company receives the material.

DOCUMENTS (2):
  • Statistical Analysis Plan (2018-02-08): https://cdn.clinicaltrials.gov/large-docs/26/NCT02564926/SAP_000.pdf
  • Study Protocol (2016-06-07): https://cdn.clinicaltrials.gov/large-docs/26/NCT02564926/Prot_001.pdf